CLINICAL TRIAL: NCT06783296
Title: Efficacy and Safety of Renal Denervation on Isolated Diastolic Hypertension: A Multicenter, Double-Blind, Randomized, Sham-Controlled Clinical Trial
Brief Title: Efficacy and Safety of Renal Denervation on Isolated Diastolic Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, professor of Medicine, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STOP
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Renal Denervation Therapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal Denervation Group (Experimental)
  Interventions: Procedure: Renal Denervation; Procedure: Renal Angiography
- Sham Control Group (Sham Comparator)
  Interventions: Procedure: Renal Angiography

INTERVENTIONS:
Procedure: Renal Denervation — Renal denervation (RDN) was performed using radiofrequency ablation in the cardiac catheterization laboratory equipped with a digital subtraction angiography (DSA) system. Under intravenous anesthesia, femoral artery access was obtained and a renal denervation sheath was advanced. An ablation catheter was then introduced to both renal arteries, and ablations were applied across four quadrants to achieve circumferential denervation. Throughout the procedure, vital signs were continuously monitored, and vasodilators or anticholinergics (e.g., nitroglycerin, atropine) were prepared to prevent vascular spasm or related complications. After completion, the femoral access site was closed and compressed, and patients were returned to the ward following stabilization of vital signs.
  Arms: Renal Denervation Group
Procedure: Renal Angiography — Renal angiography was performed under intravenous anesthesia via femoral artery access, and the procedure lasted approximately 1 hour to simulate the duration of active RDN.

SUMMARY:
This study aims to evaluate the efficacy and safety of renal denervation (RDN) in patients with isolated diastolic hypertension (IDH). The randomized, double-blind, sham-controlled, multicenter clinical trial will recruit 124 participants (62 in the treatment group and 62 in the sham control group) to assess changes in mean 24-hour ambulatory diastolic blood pressure over a 6-month follow-up period. The study is expected to provide evidence for the use of RDN as a treatment for IDH.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years, with no restriction on sex or ethnicity;
2. Diagnosis of primary hypertension, with no prior use of antihypertensive medication, and in the untreated state presenting with office systolic blood pressure (SBP) <140 mmHg and diastolic blood pressure (DBP) ≥90 mmHg, as well as 24-hour ambulatory blood pressure monitoring (ABPM) showing SBP <130 mmHg and DBP ≥80 mmHg;
3. Willingness to participate and provision of written informed consent.

Exclusion Criteria

1. DBP ≥110 mmHg;
2. Secondary hypertension;
3. Requirement for antihypertensive or blood pressure-lowering medications due to comorbid conditions (e.g., SGLT2 inhibitors, GLP-1 receptor agonists);
4. Cardiac arrhythmias interfering with blood pressure measurement (e.g., atrial fibrillation);
5. Contraindications to RDN, including renal transplantation, renal insufficiency (eGFR <45 mL/min/1.73 m²), renal artery anatomy unsuitable for the procedure (inability to access the renal vasculature; renal artery diameter <4 mm or length <20 mm; hemodynamically or anatomically significant renal artery abnormalities or stenosis; prior coronary or renal artery interventions including angioplasty or stenting), and severe hepatic impairment;
6. Contraindications to interventional procedures such as coagulopathy;
7. Pregnancy, planning pregnancy, or breastfeeding;
8. Life expectancy <1 year;
9. Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in mean 24-hour ambulatory diastolic blood pressure at 6-month follow-up | 6 months after intervention

SECONDARY OUTCOMES:
The proportion of patients achieving hypertension control without antihypertensive medication at the 6-month follow-up | 6 months after intervention
  Hypertension control without antihypertensive medication was defined as the absence of two consecutive adjudications by the Clinical Event Committee (CEC) indicating a need for oral antihypertensive therapy during the follow-up period. The CEC performed 7 adjudications throughout the study based on office blood pressure measurements obtained at biweekly visits. The CEC was blinded to treatment allocation.
Changes in 24-hour ambulatory systolic/diastolic blood pressure (daytime, nighttime, and overall periods) at the 6-month follow-up | 6 months after intervention
Changes in office systolic/diastolic blood pressure at 3, 6, and 12 months of follow-up | 3/6/12 months after intervention
Changes in home/office systolic/diastolic blood pressure at 3, 6, and 12 months of follow-up | 3/612 months after intervention
The incidence of procedure-related adverse events and complications at 6-month follow-up | 6 months after intervention
  Procedure-related adverse events and complications include renal artery stenosis, major bleeding, non-stroke thromboembolic events, renal artery stenosis or dissection, access site complications, severe vascular complications, and rehospitalization for cardiovascular events.
The incidence of major adverse cardiovascular and cerebrovascular events (MACCE) and all-cause mortality at 6-month follow-up | 6 months after intervention
  MACCE includes cardiovascular and cerebrovascular mortality, stroke, and acute heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China